CLINICAL TRIAL: NCT00005126
Title: Vietnam Era Twin (VET) Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 905
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Blood Disease; Heart Diseases; Lung Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hematologic Diseases; Heart Diseases; Lung Diseases

SUMMARY:
To conduct a baseline survey on cardiovascular, respiratory, and other major systemic disease and risk factors in members of the Vietnam Era Twin Registry.

DETAILED DESCRIPTION:
BACKGROUND:

The Vietnam Veteran Twin Registry, maintained by the NAS-NRC, was created with funding from the Veterans Administration. Department of Defense records were searched for subjects born between 1939-1957 and having the same last name and date of birth. Follow-up of induction records determined if the subjects were twins.

The registry supplemented the older World War II Veterans Twin Registry supported by the National Heart, Lung, and Blood Institute. The new registry provided an opportunity to create a resource with Black and Hispanic twins as well as whites. The new registry also included data on greater educational, socioeconomic, and lifestyle diversity than was available in the World War II Veterans Twin Registry.

DESIGN NARRATIVE:

During the first year a mailed questionnaire was designed which provided baseline data on family history, body size, morbidity, psychosocial characteristics, smoking, alcohol consumption, diet, physical activity, and drug use. The baseline data were used for analysis of cardiovascular, pulmonary, and blood diseases, and for follow-up. From the original survey, the Veterans Administration provided magnetic tape data on zygosity, smoking, alcohol consumption, heart, lung, and blood diseases, discharge rank, education, occupation, and family income. The questionnaire was completed by almost 8,900 individuals including over 3,000 twin pairs.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-04; Study Completion 1991-03 (Actual)

REFERENCES:
- [Background] Fabsitz RR, Sholinsky P, Goldberg J. Correlates of sleep problems among men: the Vietnam Era Twin Registry. J Sleep Res. 1997 Mar;6(1):50-6. doi: 10.1046/j.1365-2869.1997.00026.x. PMID 9125699